CLINICAL TRIAL: NCT04556032
Title: A Placebo-controlled, Randomized, Double-blind Trial to Assess the Effects of Ergothioneine on Cognition, Mood, and Sleep in Healthy Adult Men and Women
Brief Title: Effects of Ergothioneine on Cognition, Mood, and Sleep in Healthy Adult Men and Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated study due to unforeseen recruitment circumstances amidst the COVID19 pandemic.
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Blue California Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MB-2011
Record Dates: First submitted 2020-09-09; First posted 2020-09-21 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-Ergothioneine 10 mg/d (Experimental): Participants will receive L-Ergothioneine 10 mg capsule orally once daily for 16 weeks.
  Interventions: Dietary Supplement: L-Ergothioneine 10 mg/d
- L-Ergothioneine 25 mg/d (Experimental): Participants will receive L-Ergothioneine 25 mg capsule orally once daily for 16 weeks.
  Interventions: Dietary Supplement: L-Ergothioneine 25 mg/d
- Placebo (Placebo Comparator): Participants will receive placebo orally once daily for 16 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-Ergothioneine 10 mg/d — L-Ergothioneine 10 mg/d
  Arms: L-Ergothioneine 10 mg/d
Dietary Supplement: L-Ergothioneine 25 mg/d — L-Ergothioneine 25 mg/d
  Arms: L-Ergothioneine 25 mg/d
Other: Placebo — 0 mg/d L-Ergothioneine
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the effects of ergothioneine at two doses, compared to placebo, on cognition, mood, and sleep in healthy adult men and women.

DETAILED DESCRIPTION:
This will be a placebo-controlled, randomized, double-blind, parallel-arm trial. The study will consist of one screening (visit 1a, week 0), one baseline visit (visit 1b, week 0), and three treatment visits (visits 2, 3, and 4; weeks 4, 8, and 16).

ELIGIBILITY:
Inclusion Criteria:

* Individuals 55-79 years of age.
* Body mass index (BMI) 18.50-34.99 kg/m2
* Non-smoker defined as no smoking for at least 6 months.
* Willing to limit alcohol and caffeine consumption
* Generally, in good health based on medical history and laboratory assessments
* Agree to avoid consumption of mushrooms and excluded medications/supplements for the duration of the study
* Willing to commit to all study procedures

Exclusion Criteria:

* Consumption of mushrooms more than once per week
* History or presence of a psychiatric or neurologic disease including, but not limited to, epilepsy, cerebrovascular disturbance, traumatic injury, or clinically diagnosed dementia or Alzheimer's disease.
* Scores ≥17 on the Beck Depression Inventory
* History of cardiovascular complications, type 1 or type 2 diabetes mellitus, uncontrolled hypertension, or any other clinically significant disorder
* History of cancer except non-melanoma skin cancer or carcinoma in situ of the cervix within the past 2 years
* Use of any product containing marijuana (THC) and/or cannabidiol (CBD) including oral consumption, inhalation, & other
* Any intolerance to any components of the study products
* Exposure to any non-registered drug product within the past 30 days
* History of drug or alcohol abuse
* Considered unfit for any reason as determined by the principal investigator

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in the composite memory standard score from the Central Nervous System Vital Signs (CNS-VS) Test Battery | Baseline to Week 16

SECONDARY OUTCOMES:
Changes in the composite memory standard score from the Central Nervous System Vital Signs (CNS-VS) Test Battery | Baseline to weeks 4 and 8
Changes in standard scores for domains relating to memory, attention, and executive function from the Central Nervous System Vital Signs (CNS-VS) Test Battery | Baseline to weeks 4, 8 and 16
Changes in sleep quality based on Leeds Sleep Evaluation Questionnaire (LSEQ) | Baseline to weeks 4, 8 and 16
Changes in mood based on Profile of Mood States Questionnaire (POMS) | Baseline to weeks 4, 8 and 16

CONTACTS AND LOCATIONS:
Locations (1):
- Great Lakes Clinical Trials, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No